CLINICAL TRIAL: NCT00129129
Title: Evaluate Immuno and Safety of GSKBiologicals' HibMenCYTT vs Licensed Hib Conjugate Vaccine, Each Coadministered With Pediarix® and Prevnar®, in Healthy Infants. An Exploratory Control Group Will Receive Licensed Menomune® at 3 to 5 Years
Brief Title: Comparison of GSKBiologicals' Hib-MenCY-TT Vaccine vs Licensed Hib Conjugate or Meningococcal Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 101858; 102015 (Other: GSK)
Record Dates: First submitted 2005-08-10; First posted 2005-08-11 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2016-09

CONDITIONS: Haemophilus Influenzae Type b; Neisseria Meningitidis
Keywords: Immunogenicity; Primary & booster vaccination; Infants; Meningococcal vaccine; Safety; Children; Hib disease; Meningococcal disease
MeSH Terms: conditions — Haemophilus Infections; Meningococcal Infections | interventions — Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate; PEDIARIX; Heptavalent Pneumococcal Conjugate Vaccine; Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant

ARMS (5):
- MenHibrix Group (Experimental): Subjects in the Group were followed during the entire study period, from Day 0 up to study end 6 months post fourth dose vaccinationDuring Primary Phase (Study 101858), subjects in this group, aged 6-12 weeks at enrolment, received 3 doses of Menhibrix™ co-administered with Pediarix™ and Prevnar™ (at Day 0 and Months 2 and 4). During Fourth-Dose Phase (Study 102015), subjects primed with 3 doses of Menhibrix™ during the Primary Phase received one dose of Menhibrix™ and one concomitant dose of Prevnar™ at Month 10-13. During Primary Phase, Menhibrix™ was administered intramuscularly (IM) in the right upper thigh, and Pediarix™ and Prevnar™ IM in the left upper and lower thighs, respectively. During Fourth-Dose Phase, Menhibrix™ was administered by the same route and at the same site as during Primary Phase, and Prevnar™ was administered IM in the left upper thigh.
  Interventions: Biological: GSK Biologicals' Haemophilus influenza type b and Neisseria meningitidis serogroups C and Y-tetanus toxoid conjugate vaccine 792014 vaccine; Biological: Pediarix; Biological: Prevnar
- ActHIB Group (Active Comparator): During Primary Phase (Study 101858), subjects in this group, aged 6-12 weeks at enrolment, received 3 doses of ActHIB™ vaccine co-administered with the Pediarix™ and Prevnar™ vaccines (at Day 0 and Months 2 and 4). Subjects in this Group were followed from Day 0 up to Month 10-13 solely. During Fourth-Dose Phase (Study 102015), these subjects were followed as subjects either in the ActHIB/MenHibrix Group or in the ActHIB/ActHIB Group, receiving then one dose of either Menhibrix™ or ActHIB™ concomitantly with one dose of Prevnar™. During Primary Phase, ActHIB™ was administered intramuscularly (IM) in the right upper thigh, and the Pediarix™ and Prevnar™ vaccines IM in the left upper and lower thighs, respectively.
  Interventions: Biological: ActHIB; Biological: Pediarix; Biological: Prevnar
- Menomune Group (Active Comparator): Subjects in the Group were followed solely during the period of Primary Phase (Study 101858), up to Month 10. Subjects in the Group, aged 3-5 years at enrolment, received one dose of Menomune™ at Day 0. Menomune™ was administered subcutaneously in the left deltoid region.
  Interventions: Biological: Pediarix; Biological: Prevnar; Biological: Menomune
- ActHIB/Menhibrix Group (Experimental): Subjects in the Group were followed solely during the period of the Fourth-Dose Phase of the study (Study 102015), from Month 10-13 to Month 11-14. Subjects in this Group had been primed with ActHIB™ during Primary Phase (study 101858) and received at Month 10-13 a fourth dose of Menhibrix™ and a concomitant fourth dose of Prevnar™. Menhibrix™ and Prevnar™ were administered intramuscularly in the right and left upper thighs, respectively.
  Interventions: Biological: GSK Biologicals' Haemophilus influenza type b and Neisseria meningitidis serogroups C and Y-tetanus toxoid conjugate vaccine 792014 vaccine; Biological: ActHIB; Biological: Pediarix; Biological: Prevnar
- ActHIB/ActHIB Group (Experimental): Subjects in the Group were followed solely during the period of the Fourth-Dose Phase of the study (Study 102015), from Month 10-13 to Month 11-14. Subjects in this Group had been primed with ActHIB™ during Primary Phase of the study (study 101858) and received at Month 10-13 a fourth dose of ActHIB™ and a concomitant fourth dose of Prevnar™. ActHIB™ and Prevnar™ were administered intramuscularly in the right and left upper thighs, respectively.
  Interventions: Biological: ActHIB; Biological: Pediarix; Biological: Prevnar

INTERVENTIONS:
Biological: GSK Biologicals' Haemophilus influenza type b and Neisseria meningitidis serogroups C and Y-tetanus toxoid conjugate vaccine 792014 vaccine — Primary phase: 3 IM doses Booster phase: 1 IM dose
  Arms: ActHIB/Menhibrix Group; MenHibrix Group
Biological: ActHIB — Primary phase: 3 IM doses Booster phase: 1 IM dose
  Arms: ActHIB Group; ActHIB/ActHIB Group; ActHIB/Menhibrix Group
Biological: Pediarix — Primary phase: 3 IM doses
Biological: Prevnar — Primary phase: 3 IM doses Booster phase: 1 IM dose
Biological: Menomune — Primary phase: 1 SC dose
  Arms: Menomune Group

SUMMARY:
This study is evaluating the safety and immunogenicity of GSK Biologicals' Hib-MenCY-TT vaccine compared to a control group receiving licensed Hib conjugate vaccine, each administered at 2, 4, and 6 months of age, and compared to licensed meningococcal serogroups A, C, Y, and W-135 polysaccharide vaccine administered at 3 to 5 years of age.

The safety and immunogenicity of a booster dose of Hib-MenCY-TT vaccine will be compared to a booster dose of licensed Hib conjugate vaccine, each administered at 12 to 15 months of age. The group primed with the Hib conjugate vaccine will re-randomized at 12-15 months of age to receive a booster dose of Hib-MenCY-TT or a booster dose of the Hib conjugate vaccine.

DETAILED DESCRIPTION:
The non-inferiority of the immunogenicity, safety, and antibody persistence of Hib-MenCY-TT vaccine will be compared to ActHIB®, a monovalent Hib conjugate vaccine licensed in the US.

All subjects will be vaccinated at 2, 4, 6, and 12 to 15 months. The immunogenicity of the MenC and MenY antigens will be summarized.

MenC and MenY immunogenicity will be compared to Menomune® (a quadrivalent meningococcal A, C, Y, and W-135 plain polysaccharide vaccine licensed in the US) administered to children 3 to 5 years of age.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* For Groups A and B

  * Subjects for whom the investigator believes that parents/guardians can and will comply with the requirements of the protocol.
  * Healthy male or female between, and including, 6 and 12 weeks of age at the time of the first vaccination.
  * Written informed consent obtained from the parent or guardian of the subject.
  * Free of obvious health problems as established by medical history and clinical examination before entering the study.
  * Born after a gestation period between 36 and 42 weeks.
  * Infants who have not received a previous dose of hepatitis B vaccine or those who have received only 1 dose of hepatitis B vaccine administered at least 30 days prior to enrollment.
* For Group C

  * Subjects for whom the investigator believes that parents/guardians can and will comply with the requirements of the protocol.
  * Healthy male or female between, and including, 3 and 5 years of age at the time of the first vaccination.
  * Written informed consent obtained from the parent or guardian of the subject.
  * Free of obvious health problems as established by medical history and clinical examination before entering the study.

Exclusion Criteria:

-For Groups A and B

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of study vaccine(s).
* Previous vaccination against Neisseria meningitidis, Haemophilus influenzae type b, diphtheria, tetanus, pertussis, poliovirus, and/or Streptococcus pneumoniae; more than one previous dose of hepatitis B vaccine.
* History of Neisseria meningitidis, Haemophilus influenzae type b, diphtheria, tetanus, pertussis, hepatitis B, poliovirus, and/or Streptococcus pneumoniae disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s), including dry natural latex rubber.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at time of enrollment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

For Group C

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days of the dose of study vaccine.
* Previous vaccination against Neisseria meningitidis.
* History of Neisseria meningitidis disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, including dry natural latex rubber
* Major congenital defects or serious chronic illness.
* Acute disease at time of enrollment.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding vaccination or planned administration during the study period.

Ages: 6 Weeks to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 756 (Actual)
Dates: Start 2004-08-01; Primary Completion 2005-09-15 (Actual); Study Completion 2006-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- United States (22):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Centennial, Colorado
  - GSK Investigational Site, Norwich, Connecticut
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Bossier City, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, New Bedford, Massachusetts
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Boardman, Ohio
  - GSK Investigational Site, University Heights, Ohio
  - GSK Investigational Site, Beaver Falls, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Greenville, Pennsylvania
  - GSK Investigational Site, Norristown, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Rydal, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bryant KA, Marshall GS. Haemophilus influenzae type b-Neisseria meningitidis serogroups C and Y tetanus toxoid conjugate vaccine for infants and toddlers. Expert Rev Vaccines. 2011 Jul;10(7):941-50. doi: 10.1586/erv.11.90. PMID 21806393
- [Background] Marchant CD, Miller JM, Marshall GS, Blatter M, Aris E, Friedland LR, Boutriau D; HibMenCY-TT 005 Study Group. Randomized trial to assess immunogenicity and safety of Haemophilus influenzae type b and Neisseria meningitidis serogroups C and Y-tetanus toxoid conjugate vaccine in infants. Pediatr Infect Dis J. 2010 Jan;29(1):48-52. doi: 10.1097/INF.0b013e3181c3ce88. PMID 20035207
- [Background] Marshall GS, Marchant CD, Blatter M, Aris E, Boutriau D, Poolman JT, Friedland LR, Miller JM. Immune response and one-year antibody persistence after a fourth dose of a novel Haemophilus influenzae type b and Neisseria meningitidis serogroups C and Y-tetanus toxoid conjugate vaccine (HibMenCY) at 12 to 15 months of age. Pediatr Infect Dis J. 2010 May;29(5):469-71. doi: 10.1097/INF.0b013e3181cdd379. PMID 20072077
- [Background] Marshall GS, Marchant CD, Blatter M, Friedland LR, Aris E, Miller JM. Co-administration of a novel Haemophilus influenzae type b and Neisseria meningitidis serogroups C and Y-tetanus toxoid conjugate vaccine does not interfere with the immune response to antigens contained in infant vaccines routinely used in the United States. Hum Vaccin. 2011 Feb;7(2):258-64. doi: 10.4161/hv.7.2.14170. Epub 2011 Feb 1. PMID 21307655
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 101858 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 101858 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 101858 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 101858 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 101858 are summarised with study 102015 on the GSK Clinical Study Register.
- Available data/document: Study Protocol: 101858 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In a Primary Phase (study 101858), 3 groups, MenHibrix, ActiHIB and Menomune, were followed from Day 0 to either Month (M) 7 or 10, depending on vaccination. Then, in a Fourth-Dose Phase (study 102015), 3 groups (MenHibrix, ActiHIB/ActHIB and ActiHIB/MenHibrix) were followed from M10-13 to study end (M16-19). Treatment allocation: primary phase:
Pre-assignment Details: MenHibrix Group was followed during the entire study period, from Day 0 to M16-19). ActiHIB Group was followed as ActiHIB Group up to M10-13, when it was split into the ActHIB/ActHIB and ActHIB/MenHibrix groups, these latter being followed from M10-13 to study end. Menomune Group was followed up to M7.
Groups:
- MenHibrix Group: Subjects in the Group were followed during the entire study period, from Day 0 up to study end 6 months post fourth dose vaccination. During Primary Phase (Study 101858), subjects in this group, aged 6-12 weeks at enrolment, received 3 doses of MenHibrix™ co-administered with Pediarix™ and Prevnar™ (at Day 0 and Months 2 and 4). During Fourth-Dose Phase (Study 102015), subjects primed with 3 doses of MenHibrix™ during the Primary Phase received one dose of MenHibrix™ and one concomitant dose of Prevnar™ at Month 10-13. During Primary Phase, MenHibrix™ was administered intramuscularly (IM) in the right upper thigh, and Pediarix™ and Prevnar™ IM in the left upper and lower thighs, respectively. During Fourth-Dose Phase, MenHibrix™ was administered by the same route and at the same site as during Primary Phase, and Prevnar™ was administered IM in the left upper thigh.
- ActHIB/MenHibrix Group: Subjects primed with ActHIB vaccine who received a fourth dose of Menhibrix vaccine and a concomitant fourth dose of Prevnar vaccine during the fourth dose vaccination phase. In the fourth dose phase, Menhibrix and Prevnar vaccines were administered intramuscularly in the right and left upper thigh, respectively.
Period: Primary Phase
Arm/Group | MenHibrix Group | ActHIB Group | Menomune Group | ActHIB/MenHibrix Group | ActHIB/ActHIB Group
Started | 287 | 319 | 150 | 0 | 0
Completed | 262 | 294 | 150 | 0 | 0
Not Completed | 25 | 25 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 10 | 0 | 0 | 0
Not completed — Migration from study area | 1 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 8 | 6 | 0 | 0 | 0
Not completed — Other | 2 | 5 | 0 | 0 | 0
Period: Fourth Dose Phase
Arm/Group | MenHibrix Group | ActHIB Group | Menomune Group | ActHIB/MenHibrix Group | ActHIB/ActHIB Group
Started | 236 | 0 | 0 | 132 | 130
Completed | 232 | 0 | 0 | 128 | 124
Not Completed | 4 | 0 | 0 | 4 | 6
Not completed — Lost to Follow-up | 4 | 0 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Migration from study area | 0 | 0 | 0 | 0 | 2
Not completed — Other | 0 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MenHibrix Group | ActHIB Group | Menomune Group | Total
Number analyzed (Participants) | 287 | 319 | 150 | 756
Age, Continuous [Mean (Standard Deviation); unit: Days] | 64.2 (8.05) | 64.0 (7.52) | 1554.1 (338.4) | 560.8 (118.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 166 | 70 | 377
  Male | 146 | 153 | 80 | 379

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-polyribosyl-ribitol-phosphate (Anti-PRP) Antibody Concentration Equal to or Above (≥) Cut-off Value.
Description: The anti-PRP antibody cut-off value used for this outcome was 1.0 microgram per milliliter (µg/mL). This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: One month after the 3-dose primary vaccination course (at Month 5)
Population: The Primary According-To-Protocol (ATP) cohort for immunogenicity included all evaluable subjects (i.e. those meeting all eligibility criteria, complying with the procedures, with no elimination criteria) and for whom the data concerning the immunogenicity of at least one vaccine antigen were available during the primary phase
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 199 | 211
Participants | 186 | 181

2. Primary Outcome: Concentration of Antibodies Against Streptococcus Pneumoniae Serotypes
Description: Concentrations of antibodies are presented as geometric mean concentrations (GMCs) expressed as microgram per milliliter (µg/mL). Vaccine pneumococcal serotypes included serotypes 4, 6B, 9V, 14, 18C, 19F, 23F. This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: One month after the 3-dose primary vaccination course (at Month 5)
Population: The Primary ATP cohort for immunogenicity included all evaluable subjects (i.e. those meeting all eligibility criteria, complying with the procedures defined in the protocol, with no elimination criteria during the study) and for whom the data concerning the immunogenicity of at least one vaccine antigen were available during the primary phase.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 174 | 180
µg/mL
  Anti-4 (N=173;177) | 1.72 [1.53 to 1.94] | 1.9 [1.7 to 2.14]
  Anti-6B (N=166;162) | 1.31 [1.08 to 1.58] | 1.59 [1.35 to 1.87]
  Anti-9V (N=174;180) | 2.17 [1.93 to 2.44] | 2.32 [2.09 to 2.59]
  Anti-14 (N=167;172) | 4.79 [4.23 to 5.43] | 4.64 [4.06 to 5.31]
  Anti-18C (N=172;169) | 2.5 [2.22 to 2.83] | 2.56 [2.27 to 2.88]
  Anti-19F (N=167;169) | 1.62 [1.45 to 1.82] | 1.74 [1.57 to 1.94]
  Anti-23F (N=174;177) | 2.25 [1.92 to 2.63] | 2.46 [2.12 to 2.86]

3. Primary Outcome: Anti-pertussis Toxoid (PT), Anti-filamentous Haemagglutinin (FHA) and Anti-pertactin (PRN) Antibody Concentrations
Description: Concentrations of antibodies are presented as geometric mean concentrations (GMCs) expressed in Enzyme-Linked Immunosorbent Assay (ELISA) units per milliliter (EL.U/mL). This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: One month after the 3-dose primary vaccination course (at Month 5)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 200 | 217
EL.U/mL
  Anti-PT (N=198;215) | 57.1 [51.7 to 63.0] | 66.4 [61.0 to 72.3]
  Anti-FHA (N=200;213) | 208.9 [189.7 to 230.1] | 252.2 [228.8 to 277.9]
  Anti-PRN (N=200;217) | 86.3 [75.7 to 98.4] | 93.8 [83.1 to 105.8]

4. Primary Outcome: Number of Subjects Reporting Any Grade 3 Symptoms
Description: "Symptoms" were defined as solicited local and general symptoms and unsolicited adverse events (AEs). A "Grade 3" symptom was defined as any symptom that prevented normal everyday activity. "Any" was defined as an occurrence of any specified symptom regardless of intensity grade. This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: During the 4-day follow-up period after each primary vaccine dose
Population: The Primary Total Vaccinated cohort included all vaccinated subjects with at least one vaccine administration documented during the primary phase.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 287 | 319
Participants | 33 | 79

5. Primary Outcome: Number of Subjects With Anti-polyribosyl-ribitol-phosphate (Anti-PRP) Antibody Concentration Equal to or Above (≥) Cut-off Value
Description: The anti-PRP antibody cut-off value used for this outcome was 1.0 microgram per milliliter (µg/mL). This Outcome Measure only concerns the MenHibrix and ActHIB/ActHIB groups .
Time Frame: One month after the fourth dose (at Month 11-14)
Population: The Fourth Dose ATP cohort for immunogenicity included all evaluable subjects (i.e. those meeting eligibility criteria, complying with the procedures, with no elimination criteria) from the Fourth Dose ATP cohort for safety for whom assay results were available for antibodies 1 month (31 to 48 days) after the administration of the fourth dose.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group
Number analyzed (Participants) | 176 | 93
Participants | 174 | 92

6. Secondary Outcome: Number of Subjects With Neisseria Meningitidis Serogroup C Serum Bacterial Assay Using Rabbit Complement (rSBA-MenC) Antibody Titers ≥ the Cut-off Values
Description: rSBA-MenC antibody cut-off values for this outcome were 1:8 and 1:128.
Time Frame: Prior to and one month after the primary vaccination course (at Day 0 and Month 5 for the MenHibrix and ActHIB groups)/ prior to and one month after vaccination (at Day 0 and Month 1 for the Menomune Group)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group | Menomune Group
Number analyzed (Participants) | 177 | 194 | 136
Participants
  ≥1:8 [Prior to vaccination] (N=153;183;133) | 10 | 13 | 27
  ≥1:128 [Prior to vaccination] (N=153;183;133) | 3 | 5 | 20
  ≥1:8 [1 month post-vaccination] (N=177;194;136) | 173 | 7 | 126
  ≥1:128 [1 month post-vaccination] (N=177;194;136) | 171 | 2 | 105

7. Secondary Outcome: Neisseria Meningitidis Serogroup C Serum Bacterial Assay Using Rabbit Complement (rSBA-MenC) Antibody Titers
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenHibrix Group | ActHIB Group | Menomune Group
Number analyzed (Participants) | 177 | 194 | 136
Titers
  [Prior to vaccination] (N=153;183;133) | 4.8 [4.2 to 5.5] | 5.1 [4.4 to 5.8] | 9 [6.8 to 12.1]
  [1 month post-vaccination] (N=177;194;136) | 1096.5 [896.5 to 1341.1] | 4.4 [4.1 to 4.8] | 284.2 [210.1 to 384.3]

8. Secondary Outcome: Number of Subjects With Neisseria Meningitidis Serogroup Y Serum Bacterial Assay Using Rabbit Complement (rSBA-MenY) Antibody Titers ≥ the Cut-off Values
Description: rSBA-MenY antibody cut-off values for this outcome measure were 1:8 and 1:128.
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group | Menomune Group
Number analyzed (Participants) | 174 | 186 | 140
Participants
  ≥1:8 [Prior to vaccination] (N=156;186;140) | 29 | 28 | 92
  ≥1:128 [Prior to vaccination] (N=156;186;140) | 4 | 3 | 61
  ≥1:8 [1 month post-vaccination] (N=174;186;139) | 171 | 35 | 134
  ≥1:128 [1 month post-vaccination] (N=174;186;139) | 154 | 6 | 131

9. Secondary Outcome: Neisseria Meningitidis Serogroup Y Serum Bacterial Assay Using Rabbit Complement (rSBA-MenY) Antibody Titers
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenHibrix Group | ActHIB Group | Menomune Group
Number analyzed (Participants) | 174 | 186 | 140
Titers
  [prior to vaccination] (N=156;186;140) | 6.1 [5.2 to 7.2] | 5.7 [5.0 to 6.6] | 54.9 [38.9 to 77.5]
  [1 month post-vaccination] (N=174;186;139) | 495.3 [409.2 to 599.6] | 6.8 [5.8 to 8.1] | 685.1 [540.3 to 868.7]

10. Secondary Outcome: Number of Subjects With Neisseria Meningitidis Serogroup C Serum Bacterial Assay Using Human Complement (hSBA-MenC) Antibody Titers ≥ 1:4
Description: A composite outcome variable was formulated as follows for this immunogenicity analysis outcome: hSBA-Men titers ≥ 1:4 for subjects with post-vaccination rSBA-Men antibody titers ≥ 1:8 and lower than (<) 1:128.
Time Frame: One month after the primary vaccination course (at Month 5 for the MenHibrix and ActHIB groups)/one month after vaccination (at Month 1 for the Menomune Group)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group | Menomune Group
Number analyzed (Participants) | 177 | 22 | 136
Participants | 2 | 1 | 3

11. Secondary Outcome: Number of Subjects With Neisseria Meningitidis Serogroup Y Serum Bacterial Assay Using Human Complement (hSBA-MenC) Antibody Titers ≥ 1:4
Description: as for outcome 10
Time Frame: as for outcome 10
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group | Menomune Group
Number analyzed (Participants) | 174 | 22 | 139
Participants | 13 | 0 | 0

12. Secondary Outcome: Number of Subjects With Anti-polysaccharide C (Anti-PSC) Antibody Concentrations Above ≥ the Cut-off Values
Description: Anti-PSC antibody cut-off values for this outcome were 0.3 µg/mL and 2.0 µg/mL.
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group | Menomune Group
Number analyzed (Participants) | 197 | 207 | 138
Participants
  ≥0.3 µg/mL [prior to vaccination] (N=161;185;138) | 24 | 16 | 10
  ≥0.3 µg/mL [after vaccination] (N=197;207;136) | 196 | 8 | 134
  ≥2.0 µg/mL [prior to vaccination] (N=161;185;138) | 1 | 6 | 3
  ≥2.0 µg/mL [after vaccination] (N=197;207;136) | 172 | 0 | 122

13. Secondary Outcome: Anti-polysaccharide C (Anti-PSC) Antibody Concentrations
Description: Concentrations of antibodies are presented as geometric mean concentrations (GMCs) expressed as microgram per milliliter (µg/mL).
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | MenHibrix Group | ActHIB Group | Menomune Group
Number analyzed (Participants) | 197 | 207 | 138
µg/mL
  [prior to vaccination] (N=161;185;138) | 0.19 [0.17 to 0.21] | 0.18 [0.16 to 0.20] | 0.17 [0.16 to 0.19]
  [1 month post-vaccination] (N=197;207;136) | 4.41 [3.96 to 4.92] | 0.16 [0.15 to 0.17] | 7.37 [6.10 to 8.91]

14. Secondary Outcome: Number of Subjects With Anti-polysaccharide Y (Anti-PSY) Antibody Concentrations Equal to or Above ≥ the Cut-off Values
Description: Anti-PSY antibody cut-off values for this outcome were 0.3 µg/mL and 2.0 µg/mL.
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group | Menomune Group
Number analyzed (Participants) | 189 | 187 | 137
Participants
  ≥0.3 µg/mL [prior to vaccination] (N=157;187;137) | 23 | 28 | 6
  ≥0.3 µg/mL [after vaccination] (N=189;181;129) | 188 | 5 | 125
  ≥2.0 µg/mL [prior to vaccination] (N=157;187;137) | 5 | 6 | 2
  ≥2.0 µg/mL [after vaccination] (N=189;181;129) | 186 | 0 | 108

15. Secondary Outcome: Anti-polysaccharide Y (Anti-PSY) Antibody Concentrations
Description: as for outcome 13
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | MenHibrix Group | ActHIB Group | Menomune Group
Number analyzed (Participants) | 189 | 187 | 137
µg/mL
  [prior to vaccination] (N=157;187;137) | 0.20 [0.18 to 0.22] | 0.20 [0.18 to 0.22] | 0.17 [0.15 to 0.18]
  [1 month post-vaccination] (N=189;181;129) | 19.82 [17.40 to 22.57] | 0.15 [0.15 to 0.16] | 7.21 [5.57 to 9.34]

16. Secondary Outcome: Number of Subjects Reporting Medically Attended Visits
Description: A medically attended visit was defined as an hospitalization, an emergency room visit or a visit to or from medical personnel. This Outcome Measure only concerns subjects in the Menomune Group.
Time Frame: During the 31-day follow-up period after vaccination with Menomune vaccine at Day 0
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Menomune Group
Number analyzed (Participants) | 150
Participants
  Emergency room visit | 1
  Physician's office visit | 18

17. Secondary Outcome: Number of Subjects Reporting Rash
Description: An episode of rash was defined as an episode of hives, idiopathic thrombocytopenic purpura, petechiae. This Outcome Measure only concerns subjects in the Menomune Group.
Time Frame: During the 31-day follow-up period after vaccination with Menomune vaccine at Day 0
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Menomune Group
Number analyzed (Participants) | 150
Participants | 1

18. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject . This Outcome Measure only concerns subjects in the Menomune Group.
Time Frame: During the 31-day follow-up period after vaccination with Menomune vaccine at Day 0
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Menomune Group
Number analyzed (Participants) | 150
Participants | 0

19. Secondary Outcome: Number of Subjects With Anti-PRP Antibody Concentrations ≥ the Cut-off Values
Description: Anti-PRP antibody cut-off values for this outcome were 0.15 µg/mL and 1.0 µg/mL. This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: Prior to and one month after the primary vaccination course (at Day 0 and Month 5)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- MenHibrix Group: Subjects in the Group were followed during the entire study period from Day 0 up to study end 6 months post fourth dose vaccination. During Primary Phase (Study 101858), subjects in this group, aged 6-12 weeks at enrolment, received 3 doses of MenHibrix™ co-administered with Pediarix™ and Prevnar™ (at Day 0 and Months 2 and 4). During Fourth-Dose Phase (Study 102015), subjects primed with 3 doses of MenHibrix™ during the Primary Phase received one dose of MenHibrix™ and one concomitant dose of Prevnar™ at Month 10-13. During Primary Phase, MenHibrix™ was administered intramuscularly (IM) in the right upper thigh, and Pediarix™ and Prevnar™ IM in the left upper and lower thighs, respectively. During Fourth-Dose Phase, MenHibrix™ was administered by the same route and at the same site as during Primary Phase, and Prevnar™ was administered IM in the left upper thigh.
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 199 | 211
Participants
  ≥0.15 µg/mL [prior to vaccination] (N=112;132) | 43 | 42
  ≥0.15 µg/mL [after vaccination] (N=199;211) | 196 | 202
  ≥1.0 µg/mL [prior to vaccination] (N=112;132) | 9 | 10
  ≥1.0 µg/mL [after vaccination] (N=199;211) | 186 | 181

20. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: Concentrations of antibodies are presented as geometric mean concentrations (GMCs) expressed as microgram per milliliter (µg/mL). This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: Prior to and one month after the primary vaccination course (at Day 0 and Month 5)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 199 | 211
µg/mL
  [prior to vaccination] (N=112;132) | 0.155 [0.126 to 0.189] | 0.142 [0.117 to 0.171]
  [1 month post-vaccination] (N=199;211) | 7.992 [6.756 to 9.455] | 4.392 [3.556 to 5.425]

21. Secondary Outcome: Number of Subjects With Streptococcus Pneumoniae Serotypes Antibody Concentrations ≥ Cut-off
Description: The Streptococcus pneumoniae antibody cut-off value for this outcome was 0.05 µg/mL for the 7 serotypes in Prevnar vaccine. Prevnar vaccine pneumococcal serotypes included the serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F. This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: Prior to and one month after the primary vaccination course (at Day 0 and Month 5)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 174 | 180
Participants
  Anti-4 [prior to vaccination] (N=87;100) | 23 | 18
  Anti-4 [after vaccination] (N=173;177) | 173 | 177
  Anti-6B [prior to vaccination] (N=84;96) | 40 | 41
  Anti-6B [after vaccination] (N=166;162) | 163 | 162
  Anti-9V [prior to vaccination] (N=88;100) | 45 | 54
  Anti-9V [after vaccination] (N=174;180) | 174 | 180
  Anti-14 [prior to vaccination] (N=75;90) | 70 | 80
  Anti-14 [after vaccination] (N=167;172) | 167 | 172
  Anti-18C [prior to vaccination] (N=85;97) | 41 | 55
  Anti-18C [after vaccination] (N=172;169) | 172 | 169
  Anti-19F [prior to vaccination] (N=88;99) | 76 | 82
  Anti-19F [after vaccination] (N=167;169) | 167 | 169
  Anti-23F [prior to vaccination] (N=86;103) | 44 | 47
  Anti-23F [after vaccination] (N=174;177) | 173 | 176

22. Secondary Outcome: Number of Subjects With Streptococcus Pneumoniae Serotypes Antibody Concentrations ≥ Cut-off
Description: The Streptococcus pneumoniae antibody cut-off value for this outcome was 0.2 µg/mL for the 7 serotypes in Prevnar vaccine. Prevnar vaccine pneumococcal serotypes included the serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F. This Outcome Measure only concerns the MenHibrix and ActHIB groups
Time Frame: Prior to and one month after the primary vaccination course (at Day 0 and Month 5)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 174 | 180
Participants
  Anti-4 [prior to vaccination] (N=87;100) | 9 | 3
  Anti-4 [after vaccination] (N=173;177) | 173 | 177
  Anti-6B [prior to vaccination] (N=84;96) | 12 | 15
  Anti-6B [after vaccination] (N=166;162) | 155 | 155
  Anti-9V [prior to vaccination] (N=88;100) | 19 | 19
  Anti-9V [after vaccination] (N=174;180) | 173 | 180
  Anti-14 [prior to vaccination] (N=75;90) | 46 | 62
  Anti-14 [after vaccination] (N=167;172) | 166 | 171
  Anti-18C [prior to vaccination] (N=85;97) | 19 | 24
  Anti-18C [after vaccination] (N=172;169) | 172 | 167
  Anti-19F [prior to vaccination] (N=88;99) | 47 | 52
  Anti-19F [after vaccination] (N=167;169) | 166 | 169
  Anti-23F [prior to vaccination] (N=86;103) | 13 | 15
  Anti-23F [after vaccination] (N=174;177) | 171 | 174

23. Secondary Outcome: Number of Subjects With Streptococcus Pneumoniae Serotypes Antibody Concentrations ≥ Cut-off
Description: The Streptococcus pneumoniae antibody cut-off value for this outcome was 0.5 µg/mL for the 7 serotypes in Prevnar vaccine. Prevnar vaccine pneumococcal serotypes included the serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F. This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: Prior to and one month after the primary vaccination course (at Day 0 and Month 5)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 174 | 180
Participants
  Anti-4 [prior to vaccination] (N=87;100) | 1 | 0
  Anti-4 [after vaccination] (N=173;177) | 162 | 168
  Anti-6B [prior to vaccination] (N=84;96) | 10 | 8
  Anti-6B [after vaccination] (N=166;162) | 130 | 139
  Anti-9V [prior to vaccination] (N=88;100) | 5 | 9
  Anti-9V [after vaccination] (N=174;180) | 169 | 175
  Anti-14 [prior to vaccination] (N=75;90) | 32 | 33
  Anti-14 [after vaccination] (N=167;172) | 164 | 167
  Anti-18C [prior to vaccination] (N=85;97) | 5 | 8
  Anti-18C [after vaccination] (N=172;169) | 168 | 166
  Anti-19F [prior to vaccination] (N=88;99) | 27 | 20
  Anti-19F [after vaccination] (N=167;169) | 156 | 160
  Anti-23F [prior to vaccination] (N=86;103) | 7 | 8
  Anti-23F [after vaccination] (N=174;177) | 155 | 167

24. Secondary Outcome: Number of Subjects With Anti-diphtheria and Anti-tetanus Antibody Concentration ≥ 0.1 International Units Per Milliliter (IU/mL)
Description: The anti-diphtheria and anti-tetanus antibody cut-off value for this outcome was ≥ 0.1 IU/mL. This Outcome Measure only concerns the MenHibrix and ActHIB groups.
Time Frame: Prior to and one month after the primary vaccination course (at Day 0 and Month 5)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 201 | 220
Participants
  Anti-diphtheria [prior to vaccination] (N=118;140) | 81 | 89
  Anti-diphtheria [after vaccination] (N=201;220) | 201 | 219
  Anti-tetanus [prior to vaccination] (N=118;139) | 109 | 130
  Anti-tetanus [after vaccination] (N=199;216) | 198 | 216

25. Secondary Outcome: Anti-diphtheria and Anti-tetanus Antibody Concentrations
Description: Concentrations of antibodies are presented as geometric mean concentrations (GMCs) expressed as international units per milliliter (IU/mL). This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: Prior to and one month after the primary vaccination course (at Day 0 and Month 5)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 201 | 220
IU/mL
  Anti-diphtheria [prior to vaccination] (N=118;140) | 0.173 [0.142 to 0.210] | 0.155 [0.130 to 0.185]
  Anti-diphtheria [after vaccination] (N=201;220) | 2.060 [1.845 to 2.301] | 2.277 [2.043 to 2.537]
  Anti-tetanus [prior to vaccination] (N=118;139) | 0.565 [0.465 to 0.685] | 0.497 [0.422 to 0.585]
  Anti-tetanus [after vaccination] (N=199;216) | 3.618 [3.272 to 4.001] | 1.986 [1.773 to 2.225]

26. Secondary Outcome: Number of Subjects With Anti-hepatitis-B Surface Antigen (Anti-HBs) Antibody Concentration ≥ 10.0 Milli-international Units Per Milliliter (mIU/mL)
Description: This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: Prior to and one month after the primary vaccination course (at Day 0 and Month 5)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 171 | 169
Participants
  [prior to vaccination] (N=91;108) | 28 | 27
  [after vaccination] (N=171;169) | 167 | 166

27. Secondary Outcome: Anti-hepatitis-B Surface Antigen (Anti-HBs) Antibody Concentrations
Description: Concentrations of antibodies are presented as geometric mean concentrations (GMCs) expressed as milli-international units per milliliter (mIU/mL). This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: Prior to and one month after the primary vaccination course (at Day 0 and Month 5)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 171 | 169
mIU/mL
  [prior to vaccination] (N=91;108) | 13.5 [9.1 to 20.1] | 11.3 [8.3 to 15.4]
  [after vaccination] (N=171;169) | 1567.5 [1231.7 to 1994.9] | 1555.1 [1228 to 1969.4]

28. Secondary Outcome: Number of Subjects With Anti-PT, Anti-FHA and Anti-PRN Antibody Concentration ≥ 5.0 EL.U/mL
Description: This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: Prior to and one month after the primary vaccination course (at Day 0 and Month 5)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 200 | 217
Participants
  Anti-PT [prior to vaccination] (N=116;140) | 21 | 37
  Anti-PT [after vaccination] (N=198;215) | 196 | 214
  Anti-FHA [prior to vaccination] (N=118;140) | 91 | 103
  Anti-FHA [after vaccination] (N=200;213) | 200 | 213
  Anti-PRN [prior to vaccination] (N=117;139) | 40 | 56
  Anti-PRN [after vaccination] (N=200;217) | 199 | 215

29. Secondary Outcome: Anti PT, Anti-FHA and Anti-PRN Antibody Concentrations
Description: Concentrations of antibodies are presented as GMCs expressed as EL.U/mL. Results for one month after the 3-dose primary vaccination course (at Month 5) are presented under the Primary Outcome Measures section. This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: Prior to the primary vaccination course (at Day 0)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 118 | 140
EL.U/mL
  Anti-PT [prior to vaccination] (N=116;140) | 3.4 [3.0 to 3.8] | 3.9 [3.4 to 4.4]
  Anti-FHA [prior to vaccination] (N=118;140) | 10.0 [8.2 to 12.2] | 10.5 [8.7 to 12.8]
  Anti-PRN [prior to vaccination] (N=117;139) | 4.8 [3.9 to 5.8] | 5.1 [4.3 to 6.1]

30. Secondary Outcome: Number of Subjects With Anti-poliovirus Types 1, 2 and 3 Antibody Titer ≥ 1:8
Description: This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: Prior to and one month after the primary vaccination course (at Day 0 and Month 5)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 91 | 83
Participants
  Anti-polio 1 [prior to vaccination] (N=61;60) | 34 | 41
  Anti-polio 1 [after vaccination] (N=87;82) | 86 | 82
  Anti-polio 2 [prior to vaccination] (N=60;63) | 31 | 39
  Anti-polio 2 [after vaccination] (N=91;83) | 91 | 82
  Anti-polio 3 [prior to vaccination] (N=61;64) | 7 | 13
  Anti-polio 3 [after vaccination] (N=84;79) | 84 | 79

31. Secondary Outcome: Anti-poliovirus Types 1, 2 and 3 Antibody Titers
Description: Titers are presented as geometric mean titers (GMTs). This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: Prior to and one month after the primary vaccination course (at Day 0 and Month 5)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 91 | 83
Titers
  Anti-polio 1 [prior to vaccination] (N=61;60) | 12.3 [8.8 to 17.2] | 17.3 [12.4 to 24.2]
  Anti-polio 1 [after vaccination] (N=87;82) | 530.7 [409.7 to 687.5] | 651.5 [501.7 to 846.0]
  Anti-polio 2 [prior to vaccination] (N=60;63) | 9.4 [7.1 to 12.3] | 13.5 [9.9 to 18.5]
  Anti-polio 2 [after vaccination] (N=91;83) | 398.2 [304.7 to 520.3] | 330.4 [242.8 to 449.6]
  Anti-polio 3 [prior to vaccination] (N=61;64) | 4.7 [4.1 to 5.2] | 6.2 [4.7 to 8.2]
  Anti-polio 3 [after vaccination] (N=84;79) | 923.7 [696.1 to 1225.8] | 1055.8 [813.4 to 1370.5]

32. Secondary Outcome: Number of Subjects With Vaccine Response to PT, FHA and PRN
Description: Vaccine response to PT/FHA/PRN was defined as, for initially seronegative subjects, antibody concentration ≥ 5 EL.U/mL one month post-primary vaccination course, and, for initially seropositive subjects, antibody concentration one month post-primary vaccination course ≥ 1-fold the pre-vaccination antibody concentration. A seronegative/seronegative subject was defined as a subject with antibody concentration </≥ 5 EL.U/mL for anti-PT/FHA/PRN prior to vaccination. This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: One month after the 3-dose primary vaccination course (at Month 5)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 116 | 135
Participants
  Anti-PT (N=111;135) | 109 | 132
  Anti-FHA (N=116;132) | 113 | 128
  Anti-PRN (N=115;133) | 103 | 126

33. Secondary Outcome: Number of Subjects Reporting Any, Grade 2 or 3 and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms were pain, redness and swelling at injection site. "Any" = any report of the specified symptom irrespective of intensity grade; "Grade 2 pain" = cried/protested on touch; "Grade 3 pain" = cried when limb was moved/spontaneously painful; "Grade 2 or 3" redness/swelling = redness/swelling larger than (>) 10 millimeters (mm); "Grade 3" redness/swelling = redness/swelling > 30 mm. This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: Within 4 days (Day 0-3) after the 3-dose primary vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 286 | 317
Participants
  Any pain | 129 | 171
  Grade 2 or 3 pain | 62 | 90
  Grade 3 pain | 13 | 31
  Any redness | 112 | 148
  Redness >10 mm | 22 | 31
  Redness >30 mm | 1 | 11
  Any swelling | 90 | 110
  Swelling >10 mm | 27 | 27
  Swelling >30 mm | 1 | 11

34. Secondary Outcome: Number of Subjects Reporting Any, Grade 2 or 3 and Grade 3 Solicited Local Symptoms
Description: as for outcome 33
Time Frame: Within 8 days (Day 0-7) after the 3-dose primary vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 286 | 317
Participants
  Any pain | 129 | 171
  Grade 2 or 3 pain | 63 | 90
  Grade 3 pain | 13 | 31
  Any redness | 113 | 148
  Redness >10 mm | 22 | 31
  Redness >30 mm | 1 | 11
  Any swelling | 90 | 111
  Swelling >10 mm | 27 | 27
  Swelling >30 mm | 1 | 11

35. Secondary Outcome: Number of Subjects Reporting Any, Grade 2 or 3 and Grade 3 Solicited General Symptoms
Description: Solicited general symptoms were fever, irritability/fussiness, drowsiness, and loss of appetite. "Any" = any report of the specified symptom irrespective of intensity grade and relationship to vaccination. "Grade 2" for Drowsiness, Irritability/Fussiness and Loss of appetite = symptom that interfered with normal activity; "Grade 3" for Drowsiness and Irritability/Fussiness = symptom that prevented normal activity; "Grade 3" Loss of appetite = not eating at all. Fever = rectal temperature ≥ 38.0 degrees Celsius (°C); "Grade 2 or 3" fever = rectal temperature higher than (>) 39°C; "Grade 3" fever = rectal temperature > 40°C. This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: Within 4 days (Day 0-3) after the 3-dose primary vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 286 | 317
Participants
  Any drowsiness | 185 | 224
  Grade 2 or 3 drowsiness | 84 | 112
  Grade 3 drowsiness | 9 | 20
  Fever ≥38.0°C | 110 | 150
  Fever >39.0°C | 14 | 13
  Fever >40.0°C | 0 | 0
  Any irritability | 217 | 268
  Grade 2 or 3 irritability | 125 | 161
  Grade 3 irritability | 22 | 48
  Any loss of appetite | 123 | 159
  Grade 2 or 3 loss of appetite | 32 | 51
  Grade 3 loss of appetite | 3 | 4

36. Secondary Outcome: Number of Subjects Reporting Any, Grade 2 or 3 and Grade 3 Solicited General Symptoms
Description: Solicited general symptoms were fever, irritability/fussiness, drowsiness, and loss of appetite. "Any" = any report of the specified symptom irrespective of intensity grade and relationship to vaccination. "Grade 2" for Drowsiness, Irritability/Fussiness and Loss of appetite = symptom that interfered with normal activity; "Grade 3" for Drowsiness and Irritability/Fussiness = symptom that prevented normal activity; "Grade 3" Loss of appetite = not eating at all. Fever = rectal temperature ≥ 38.0 degrees Celsius (°C); "Grade 2 or 3" fever = rectal temperature higher than (>) 39°C; "Grade 3" fever = rectal temperature > 40°C. This Outcome Measure only concerns the MenHibrix and ActHIB groups
Time Frame: Within 8 days (Day 0-7) after the 3-dose primary vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 286 | 317
Participants
  Any drowsiness | 187 | 227
  Grade 2 or 3 drowsiness | 85 | 116
  Grade 3 drowsiness | 10 | 21
  Fever ≥38.0°C | 115 | 158
  Fever >39.0°C | 19 | 19
  Fever >40.0°C | 0 | 0
  Any irritability | 222 | 272
  Grade 2 or 3 irritability | 127 | 168
  Grade 3 irritability | 25 | 51
  Any loss of appetite | 127 | 164
  Grade 2 or 3 loss of appetite | 35 | 56
  Grade 3 loss of appetite | 4 | 5

37. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: From Dose 1 (at Day 0) through Day 30 following the last vaccine dose administered (Day 30 post Month 4 vaccination for MenHibrix and ActHIB groups, Day 30 post Month 1 for Menomune Group).
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group | Menomune Group
Number analyzed (Participants) | 287 | 319 | 150
Participants | 213 | 230 | 37

38. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: During the entire Primary Phase of the study, from Day 0 up to the end of Primary Phase safety follow-up period (6 months after the last vaccination).
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group | Menomune Group
Number analyzed (Participants) | 287 | 319 | 150
Participants | 16 | 20 | 0

39. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects. This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: From Day 0 following Dose 1 throughout the study up to the day preceding the administration of the fourth dose of vaccine.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 287 | 319
Participants | 16 | 20

40. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Illness(es) (NOCIs)
Description: NOCIs include autoimmune disorders, asthma, type I diabetes, allergies. This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: as for outcome 39
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 287 | 319
Participants | 2 | 5

41. Secondary Outcome: Number of Subjects Reporting Rash
Description: An episode of rash was defined as an episode of hives, idiopathic thrombocytopenic purpura, petechiae. This Outcome Measure only concerns the MenHibrix and ActHIB groups .
Time Frame: as for outcome 39
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 287 | 319
Participants | 50 | 55

42. Secondary Outcome: Number of Subjects Reporting Emergency Room (ER) Visits or Visits to Physicians' Office, Related or Not to Common Illnesses
Description: Emergency room (ER) visits or physicians office visits assessed were those unrelated to well-child care, vaccination, injury or common acute illnesses such as upper respiratory tract infections, otitis media, pharyngitis, gastroenteritis. This Outcome Measure only concerns the MenHibrix and ActHIB groups.
Time Frame: as for outcome 39
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB Group
Number analyzed (Participants) | 287 | 319
Participants
  Emergency room visit | 25 | 31
  Physician's office visit | 181 | 190
  Physician's o. v. not related to common illnesses | 51 | 46

43. Secondary Outcome: Number of Subjects With Fourth Dose Response for Neisseria Meningitidis Serogroup C and Y Serum Bacterial Assay Using Rabbit Complement (rSBA-MenC and Y)
Description: Fourth dose responses to rSBA-MenC and rSBA-MenY were defined as follows (Definition 1):
  * Initially seronegative subjects (pre-fourth dose antibody titer below cut-off: < 1:8) should have an antibody titer at least four-fold higher than the cut-off, one month after fourth dose (post-fourth dose antibody titer ≥1:32),
  * Initially seropositive subjects (pre-fourth dose antibody titer above cut-off: ≥1:8) should have an antibody titer at least four-fold higher than the pre-fourth dose antibody titer, one month after fourth dose.
Time Frame: One month post fourth dose vaccination (at Month 11-14)
Population: The Fourth Dose ATP cohort for immunogenicity included evaluable subjects (i.e. those meeting eligibility criteria, complying with the procedures, with no elimination criteria) from the Fourth Dose ATP cohort for safety for whom assay results were available for antibodies against study vaccine antigen at 31 to 48 days post fourth dose vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- ActHIB/ActHIB Group: Subjects in the Group were followed solely during the period of the Fourth-Dose Phase of the study (Study 102015), from Month 10-13 to Month 11-14. Subjects in this Group had been primed with ActHIB™ during Primary Phase (study 101858) and received at Month 10-13 a fourth dose of MenHibrix™ and a concomitant fourth dose of Prevnar™. MenHibrix™ and Prevnar™ were administered intramuscularly in the right and left upper thighs, respectively.
- ActHIB/MenHibrix Group: Subjects in the Group were followed solely during the period of the Fourth-Dose Phase of the study (Study 102015), from Month 10-13 to Month 11-14. Subjects in this Group had been primed with ActHIB™ during Primary Phase of the study (study 101858) and received at Month 10-13 a fourth dose of ActHIB™ and a concomitant fourth dose of Prevnar™. ActHIB™ and Prevnar™ were administered intramuscularly in the right and left upper thighs, respectively.
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 149 | 72 | 79
Participants
  rSBA-MenC (N=149;72;77) | 131 | 2 | 71
  rSBA-MenY (N=147;67;79) | 119 | 10 | 76

44. Secondary Outcome: Number of Subjects With Fourth Dose Response for Neisseria Meningitidis Serogroup C and Y Serum Bacterial Assay Using Rabbit Complement (rSBA-MenC and Y)
Description: Fourth dose responses to rSBA-MenC and rSBA-MenY were also assessed using a second definition (Definition 2):
  * Post-fourth dose rSBA antibody titers ≥1:32 in subjects seronegative at the pre-fourth dose time point (rSBA antibody titers < 1:8),
  * At least (i.e., greater than or equal to) a 4-fold rise in rSBA antibody titers in subjects with pre-fourth dose antibody titers ≥1:8 but < 1:128,
  * At least (i.e., greater than or equal to) a 2-fold rise in rSBA antibody titers in subjects with pre-fourth dose antibody titers ≥1:128.
Time Frame: One month post fourth dose vaccination (at Month 11-14)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 149 | 72 | 79
Participants
  rSBA-MenC (N=149;72;77) | 140 | 2 | 71
  rSBA-MenY (N=147;67;79) | 134 | 11 | 78

45. Secondary Outcome: Number of Subjects With Fourth Dose Response for Neisseria Meningitidis Serogroup C and Y Serum Bacterial Assay Using Human Complement (hSBA-MenC and Y)
Description: Fourth dose responses to hSBA-MenC and hSBA-MenY were defined as follows (Definition 1):
  * Initially seronegative subjects (pre-fourth dose antibody titer below cut-off: < 1:8) should have an antibody titer at least four-fold higher than the cut-off, one month after the fourth dose (post-fourth dose antibody titer ≥1:16),
  * Initially seropositive subjects (pre-fourth dose antibody titer above cut-off: ≥1:8) should have an antibody titer at least four-fold higher than the pre-fourth dose antibody titer, one month after the fourth dose.
Time Frame: One month post fourth dose vaccination (at Month 11-14)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Groups:
- Menhibrix Group: Subjects of 6-12 weeks of age received 3 doses of Menhibrix vaccine co-administered with Pediarix and Prevnar vaccines during the primary vaccination phase. Subjects received a fourth dose of Menhibrix vaccine and a concomitant fourth dose of Prevnar vaccine during the fourth dose vaccination phase. In the primary phase, Menhibrix vaccine was administered intramuscularly into the right upper thigh. Pediarix and Prevnar vaccines were administered intramuscularly into the left upper thigh and the left lower thigh, respectively. In the fourth dose phase, Menhibrix vaccine was administered by the same route at the same vaccination site and Prevnar was administered intramuscularly in the left upper thigh.
Arm/Group | Menhibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 61 | 36 | 33
Participants
  hSBA-MenC (N=58;36;33) | 44 | 0 | 29
  hSBA-MenY (N=61;36;33) | 52 | 1 | 15

46. Secondary Outcome: Number of Subjects With Fourth Dose Response for Neisseria Meningitidis Serogroup C and Y Serum Bacterial Assay Using Human Complement (hSBA-MenC and Y)
Description: Fourth dose responses to hSBA-MenC and hSBA-MenY were also assessed using a second definition (Definition 2):
  * Post-fourth dose hSBA antibody titers ≥1:16 in subjects seronegative at the pre-fourth dose time point (hSBA antibody titers < 1:8),
  * At least (i.e., greater than or equal to) a 4-fold rise in hSBA antibody titers in subjects with pre-fourth dose antibody titers ≥1:4 but < 1: 8,
  * At least (i.e., greater than or equal to) a 2-fold rise in hSBA antibody titers in subjects with pre-fourth dose antibody titers ≥1:8.
Time Frame: One month post fourth dose vaccination (at Month 11-14)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 61 | 36 | 33
Participants
  hSBA-MenC (N=58;36;33) | 52 | 0 | 29
  hSBA-MenY (N=61;36;33) | 56 | 1 | 15

47. Secondary Outcome: Number of Subjects With Streptococcus Pneumoniae Serotypes Antibody Concentrations Equal to or Above 0.05 Microgram Per Milliliter (µg/mL)
Description: Streptococcus pneumoniae antibody cut-off values assessed was ≥0.05 µg/mL for the 7 serotypes in Prevnar vaccine.
  Vaccine pneumococcal serotypes included serotypes 4, 6B, 9V, 14, 18C, 19F, 23F.
Time Frame: One month after fourth dose vaccination (at Month 11-14)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 176 | 90 | 102
Participants
  Anti-4 (N=174;89;102) | 174 | 89 | 102
  Anti-6B (N=174;89;101) | 174 | 89 | 101
  Anti-9V (N=175;90;102) | 175 | 90 | 102
  Anti-14 (N=174;87;100) | 174 | 87 | 100
  Anti-18C (N=175;88;102) | 175 | 88 | 102
  Anti-19F (N=173;89;96) | 173 | 89 | 96
  Anti-23F (N=176;90;102) | 175 | 90 | 101

48. Secondary Outcome: Number of Subjects With Streptococcus Pneumoniae Serotypes Antibody Concentrations Equal to or Above 0.2 Microgram Per Milliliter (µg/mL)
Description: Streptococcus pneumoniae antibody cut-off values assessed was ≥0.2 µg/mL for the 7 serotypes in Prevnar vaccine.
  Vaccine pneumococcal serotypes included serotypes 4, 6B, 9V, 14, 18C, 19F, 23F.
Time Frame: One month after fourth dose vaccination (at Month 11-14)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 176 | 90 | 102
Participants
  Anti-4 (N=174;89;102) | 174 | 89 | 102
  Anti-6B (N=174;89;101) | 174 | 89 | 101
  Anti-9V (N=175;90;102) | 175 | 90 | 102
  Anti-14 (N=174;87;100) | 174 | 87 | 100
  Anti-18C (N=175;88;102) | 175 | 88 | 102
  Anti-19F (N=173;89;96) | 171 | 89 | 96
  Anti-23F (N=176;90;102) | 175 | 90 | 101

49. Secondary Outcome: Number of Subjects With Streptococcus Pneumoniae Serotypes Antibody Concentrations Equal to or Above 0.5 Microgram Per Milliliter (µg/mL)
Description: Streptococcus pneumoniae antibody cut-off values assessed was ≥0.5 µg/mL for the 7 serotypes in Prevnar vaccine.
  Vaccine pneumococcal serotypes included serotypes 4, 6B, 9V, 14, 18C, 19F, 23F.
Time Frame: One month after fourth dose vaccination (at Month 11-14)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 176 | 90 | 102
Participants
  Anti-4 (N=174;89;102) | 165 | 86 | 99
  Anti-6B (N=174;89;101) | 171 | 89 | 100
  Anti-9V (N=175;90;102) | 174 | 90 | 102
  Anti-14 (N=174;87;100) | 172 | 87 | 100
  Anti-18C (N=175;88;102) | 174 | 88 | 102
  Anti-19F (N=173;89;96) | 157 | 83 | 91
  Anti-23F (N=176;90;102) | 175 | 90 | 101

50. Secondary Outcome: Concentration of Antibodies Against Streptococcus Pneumonia Serotypes
Description: Concentrations of antibodies are presented as geometric mean concentrations (GMCs) expressed as microgram per milliliter (µg/mL).
  Vaccine pneumococcal serotypes included serotypes 4, 6B, 9V, 14, 18C, 19F, 23F.
Time Frame: One month post fourth dose vaccination (at Month 11-14)
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Menhibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 176 | 90 | 102
µg/mL
  Anti-4 (N=174;89;102) | 2.38 [2.10 to 2.70] | 2.69 [2.26 to 3.21] | 2.92 [2.46 to 3.48]
  Anti-6B (N=174;89;101) | 3.91 [3.45 to 4.44] | 4.07 [3.37 to 4.90] | 5.04 [4.30 to 5.92]
  Anti-9V (N=175;90;102) | 3.84 [3.42 to 4.31] | 3.85 [3.25 to 4.56] | 4.60 [3.93 to 5.38]
  Anti-14 (N=174;87;100) | 6.12 [5.39 to 6.94] | 7.00 [5.97 to 8.19] | 7.87 [6.75 to 9.19]
  Anti-18C (N=175;88;102) | 4.57 [3.99 to 5.24] | 5.23 [4.46 to 6.12] | 5.45 [4.50 to 6.58]
  Anti-19F (N=173;89;96) | 1.81 [1.56 to 2.09] | 1.93 [1.60 to 2.33] | 2.04 [1.73 to 2.41]
  Anti-23F (N=176;90;102) | 7.23 [6.21 to 8.41] | 8.02 [6.65 to 9.68] | 9.08 [7.25 to 11.38]

51. Secondary Outcome: Number of Subjects With Anti-polyribosyl-ribitol-phosphate (Anti-PRP) Antibody Concentrations Equal to or Above the Cut-off Values
Description: Anti-PRP antibody cut-off values assessed were ≥0.15 µg/mL and ≥1.0 µg/mL.
Time Frame: Prior to and one month after the fourth dose (at Month 10-13 and at Month 11-14)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 176 | 93 | 103
Participants
  ≥0.15 µg/mL [pre-4th dose] (N=160;89;95) | 152 | 78 | 85
  ≥0.15 µg/mL [post-4th dose] (N=176;93;103) | 176 | 93 | 103
  ≥1.0 µg/mL [pre-4th dose] (N=160;89;95) | 90 | 41 | 40
  ≥1.0 µg/mL [post-4th dose] (N=176;93;103) | 174 | 92 | 101

52. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: as for outcome 13
Time Frame: Prior to and one month after the fourth dose (at Month 10-13 and at Month 11-14)
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/Menhibrix Group
Number analyzed (Participants) | 176 | 93 | 103
µg/mL
  [pre-fourth dose] (N=160;89;95) | 1.073 [0.897 to 1.284] | 0.810 [0.599 to 15095] | 0.695 [0.520 to 0.928]
  [post-fourth dose] (N=176;93;103) | 28.596 [24.300 to 33.652] | 19.029 [14.895 to 24.311] | 10.650 [8.520 to 13.314]

53. Secondary Outcome: Number of Subjects With Neisseria Meningitidis Serogroup C Serum Bacterial Assay Using Rabbit Complement (rSBA-MenC) Antibody Titers Equal to or Above the Cut-off Values
Description: rSBA-MenC antibody cut-off values assessed were ≥1:8 and ≥1:128
Time Frame: Prior to and one month after the fourth dose (at Month 10-13 and at Month 11-14)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | Menhibrix Group | ActHIB/ActHIB Group | ActHIB/Menhibrix Group
Number analyzed (Participants) | 163 | 83 | 92
Participants
  ≥ 1:8 [pre-fourth dose] (N=157;83;89) | 147 | 5 | 9
  ≥1:8 [post-fourth dose] (N=163;82;92) | 161 | 8 | 90
  ≥ 1:128 [pre-fourth dose] (N=157;83;89) | 104 | 1 | 2
  ≥1:128 [post-fourth dose] (N=163;82;92) | 159 | 1 | 74

54. Secondary Outcome: rSBA-MenC Antibody Titers
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: Prior to and one month after the fourth dose (at Month 10-13 and at Month 11-14)
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 163 | 83 | 92
Titers
  [pre-fourth dose] (N=157;83;89) | 167.1 [134.1 to 208.2] | 4.7 [4.1 to 5.5] | 5.3 [4.4 to 6.4]
  [post-fourth dose] (N=163;82;92)) | 2443.9 [1981.1 to 3014.7] | 5.3 [4.3 to 6.5] | 321.8 [246.8 to 419.5]

55. Secondary Outcome: Number of Subjects With Neisseria Meningitidis Serogroup Y Serum Bacterial Assay Using Rabbit Complement (rSBA-MenY) Antibody Titers Equal to or Above the Cut-off Values
Description: rSBA-MenY antibody cut-off values assesse were ≥1:8 and ≥1:128.
Time Frame: Prior to and one month after the fourth dose (at Month 10-13 and at Month 11-14)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 162 | 80 | 93
Participants
  ≥1:8 [pre-fourth dose] (N=158;79;90) | 142 | 26 | 37
  ≥1:8 [post-fourth dose] (N=162;80;93) | 160 | 30 | 93
  ≥1:128 [pre-fourth dose] (N=158;79;90) | 96 | 10 | 17
  ≥1:128 [post-fourth dose] (N=162;80;93) | 158 | 16 | 92

56. Secondary Outcome: rSBA-MenY Antibody Titers
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: Prior to and one month after the fourth dose (at Month 10-13 and at Month 11-14)
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 162 | 80 | 93
Titers
  [pre-fourth dose] (N=158;79;90) | 128.6 [101.2 to 163.5] | 11.3 [7.9 to 16.1] | 15.6 [10.7 to 22.7]
  [post-fourth dose] (N=162;80;93) | 1424.6 [1187.8 to 1708.8] | 16.1 [10.5 to 24.6] | 1454.0 [1151.5 to 1836.1]

57. Secondary Outcome: Number of Subjects With Neisseria Meningitidis Serogroup C Serum Bacterial Assay Using Human Complement (hSBA-MenC) Antibody Titers Equal to or Above the Cut-off Values
Description: hSBA-MenC antibody cut-off values assessed were ≥1:4 and ≥1:8.
Time Frame: Prior to and one month after the fourth dose (at Month 10-13 and at Month 11-14)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 65 | 38 | 35
Participants
  ≥1:4 [pre-fourth dose] (N=59;38;35) | 54 | 0 | 1
  ≥1:4 [post-fourth dose] (N=65;37;35) | 63 | 1 | 33
  ≥1:8 [pre-fourth dose] (N=59;38;35) | 54 | 0 | 0
  ≥1:8 [post-fourth dose] (N=65;37;35) | 63 | 0 | 33

58. Secondary Outcome: hSBA-MenC Antibody Titers
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: Prior to and one month after the fourth dose (at Month 10-13 and at Month 11-14)
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 65 | 38 | 35
Titers
  [pre-fourth dose] (N=59;38;35) | 68.1 [46.1 to 100.7] | NA [NA to NA] — Not calculable as no subject had hSBA-MenY titers equal to or above the assay cut-off values. | 2.0 [2.0 to 2.1]
  [post-fourth dose] (N=65;37;35) | 657.1 [438.4 to 984.8] | 2.1 [1.9 to 2.2] | 72.5 [46.4 to 113.3]

59. Secondary Outcome: Number of Subjects With Neisseria Meningitidis Serogroup Y Serum Bacterial Assay Using Human Complement (hSBA-MenY) Antibody Titers Equal to or Above the Cut-off Values
Description: hSBA-MenY antibody cut-off values assessed were ≥1:4 and ≥1:8.
Time Frame: Prior to and one month after the fourth dose (at Month 10-13 and at Month 11-14)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 65 | 38 | 35
Participants
  ≥1:4 [pre-fourth dose] (N=62;38;35) | 33 | 0 | 0
  ≥1:4 [post-fourth dose] (N=65;37;35) | 62 | 1 | 21
  ≥1:8 [pre-fourth dose] (N=62;38;35) | 30 | 0 | 0
  ≥1:8 [post-fourth dose] (N=65;37;35) | 62 | 1 | 20

60. Secondary Outcome: hSBA-MenY Antibody Titers
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: Prior to and one month after the fourth dose (at Month 10-13 and at Month 11-14)
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 65 | 38 | 35
Titers
  [pre-fourth dose] (N=62;38;35) | 11.3 [7.1 to 18.0] | NA [NA to NA] — Not calculable as no subject had hSBA-MenY titers equal to or above the assay cut-off values. | NA [NA to NA] — Not calculable as no subject had hSBA-MenY titers equal to or above the assay cut-off values.
  [post-fourth dose] (N=65;37;35) | 246.6 [168.0 to 362.1] | 2.2 [1.8 to 2.6] | 11.1 [6.5 to 19.0]

61. Secondary Outcome: Number of Subjects With Anti-polysaccharide C (Anti-PSC) Antibody Concentrations Equal to or Above the Cut-off Values
Description: Anti-PSC antibody cut-off values assessed were ≥0.3 µg/mL and ≥2.0 µg/mL.
Time Frame: Prior to and one month after the fourth dose (at Month 10-13 and at Month 11-14)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 174 | 89 | 104
Participants
  ≥0.3 µg/mL [pre-fourth dose] (N=159;89;89) | 150 | 3 | 5
  ≥0.3 µg/mL [post-fourth dose] (N=174;89;104) | 173 | 3 | 104
  ≥2.0 µg/mL [pre-fourth dose] (N=159;89;89) | 20 | 0 | 1
  ≥2.0 µg/mL [post-fourth dose] (N=174;89;104) | 142 | 0 | 98

62. Secondary Outcome: Anti-PSC Antibody Concentrations
Description: as for outcome 13
Time Frame: Prior to and one month after the fourth dose (at Month 10-13 and at Month 11-14)
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 174 | 89 | 104
µg/mL
  [pre-fourth dose] (N=159;89;89) | 0.88 [0.77 to 1.00] | 0.16 [0.15 to 0.16] | 0.16 [0.15 to 0.18]
  [post-fourth dose] (N=174;89;104) | 4.32 [3.77 to 4.95] | 0.16 [0.15 to 0.16] | 6.81 [5.84 to 7.95]

63. Secondary Outcome: Number of Subjects With Anti-polysaccharide Y (Anti-PSY) Antibody Concentrations Equal to or Above the Cut-off Values
Description: Anti-PSY antibody cut-off values assessed were ≥0.3 µg/mL and ≥2.0 µg/mL.
Time Frame: Prior to and one month after the fourth dose (at Month 10-13 and at Month 11-14)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 173 | 87 | 101
Participants
  ≥0.3 µg/mL [pre-fourth dose] (N=157;82;85) | 155 | 1 | 0
  ≥0.3 µg/mL [post-fourth dose] (N=173;87;101) | 172 | 3 | 101
  ≥2.0 µg/mL [pre-fourth dose] (N=157;82;85) | 116 | 0 | 0
  ≥2.0 µg/mL [post-fourth dose] (N=173;87;101) | 168 | 0 | 87

64. Secondary Outcome: Anti-PSY Antibody Concentrations
Description: as for outcome 13
Time Frame: Prior to and one month after the fourth dose (at Month 10-13 and at Month 11-14)
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 173 | 87 | 101
µg/mL
  [pre-fourth dose] (N=157;82;85) | 3.83 [3.27 to 4.48] | 0.15 [0.15 to 0.16] | NA [NA to NA] — Not calculable as no subject had anti-PSY antibody concentration equal to or above the assay cut-off values.
  [post-fourth dose] (N=173;87;101) | 22.27 [19.04 to 26.04] | 0.16 [0.15 to 0.16] | 5.57 [4.66 to 6.64]

65. Secondary Outcome: Number of Subjects With Anti-tetanus Antibody Concentration Equal to or Above 0.1 International Units Per Milliliter (IU/mL)
Time Frame: Prior to and one month after the fourth dose (at Month 10-13 and at Month 11-14)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 178 | 95 | 104
Participants
  [pre-fourth dose] (N=164;92;95) | 164 | 89 | 93
  [post-fourth dose] (N=178;95;104) | 178 | 95 | 104

66. Secondary Outcome: Anti-tetanus Antibody Concentrations
Description: Concentrations of antibodies are presented as geometric mean concentrations (GMCs) expressed as international units per milliliter (IU/mL).
Time Frame: Prior to and one month after the fourth dose (at Month 10-13 and at Month 11-14)
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 178 | 95 | 104
IU/mL
  [pre-fourth dose] (N=164;92;95) | 0.782 [0.711 to 0.861] | 0.461 [0.384 to 0.554] | 0.488 [0.409 to 0.582]
  [post-fourth dose] (N=178;95;104) | 2.559 [2.333 to 2.806] | 1.785 [1.484 to 2.147] | 1.794 [1.474 to 2.184]

67. Secondary Outcome: Number of Subjects Reporting Any, Grade 2 or 3 and Grade 3 Solicited Local Symptoms
Description: Solicited symptoms assessed were pain, redness, swelling at the injection site and increase in limb circumference. "Any"= any report of the specified symptom irrespective of intensity grade; "Grade 2 pain" = cried/protested on touch; "Grade 3 pain" = cried when limb was moved/spontaneously painful; "Grade 2 or 3" redness/swelling = redness/swelling >10 millimeters (mm); "Grade 3" redness/swelling = redness/swelling >30 mm; "Grade 2" limb circumference (LC) = LC >20 mm; "Grade 3" LC = LC >40 mm
Time Frame: Within 4 days (Day 0-3) after fourth dose vaccination
Population: The Fourth Dose Total Vaccinated cohort included all vaccinated subjects during the fourth dose phase
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 232 | 126 | 130
Participants
  Any limb circumference | 59 | 44 | 36
  Limb circumference >20 mm | 2 | 5 | 5
  Limb circumference >40 mm | 0 | 0 | 0
  Any pain | 79 | 42 | 48
  Grade 2 or 3 pain | 26 | 15 | 12
  Grade 3 pain | 3 | 2 | 3
  Any redness | 81 | 40 | 38
  Redness >10 mm | 12 | 10 | 10
  Redness >30 mm | 4 | 3 | 3
  Any swelling | 49 | 19 | 20
  Swelling >10 mm | 9 | 1 | 6
  Swelling >30 mm | 3 | 0 | 0

68. Secondary Outcome: Number of Subjects Reporting Any, Grade 2 or 3 and Grade 3 Solicited Local Symptoms
Description: as for outcome 67
Time Frame: Within 8 days (Day 0-7) after fourth dose vaccination
Population: The Fourth Dose Total Vaccinated cohort included all vaccinated subjects during the fourth dose phase.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 232 | 126 | 130
Participants
  Any limb circumference | 61 | 46 | 36
  Limb circumference >20 mm | 2 | 5 | 5
  Limb circumference >40 mm | 0 | 0 | 0
  Any pain | 79 | 42 | 48
  Grade 2 or 3 pain | 26 | 15 | 12
  Grade 3 pain | 3 | 2 | 3
  Any redness | 81 | 40 | 39
  Redness >10 mm | 12 | 10 | 11
  Redness >30 mm | 4 | 3 | 4
  Any swelling | 49 | 19 | 20
  Swelling > 10 mm | 9 | 1 | 6
  Swelling > 30 mm | 3 | 0 | 0

69. Secondary Outcome: Number of Subjects Reporting Any, Grade 2 or 3 and Grade 3 Solicited General Symptoms
Description: Solicited general symptoms assessed were fever, irritability/fussiness, drowsiness, loss of appetite. "Any"= any report of the specified symptom irrespective of intensity and relationship to vaccination. "Grade 2" for Drowsiness, Irritability/Fussiness & Loss of appetite = interfered with normal activity; "Grade 3" for Drowsiness, Irritability/Fussiness = prevented normal activity; "Grade 3" Loss of appetite = not eating at all; Fever = rectal temperature (T) ≥38.0 degrees Celsius (°C); "Grade 2 or 3" for fever = T >39.0°C; "Grade 3" for fever = T >40.0°C
Time Frame: Within 4 days (Day 0-3) after fourth dose vaccination
Population: The Fourth Dose Total Vaccinated cohort included all vaccinated subjects during the fourth dose phase.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 232 | 126 | 130
Participants
  Any drowsinnes | 72 | 48 | 41
  Grade 2 or 3 drowsiness | 21 | 7 | 7
  Grade 3 drowsiness | 2 | 1 | 1
  Fever ≥ 38.0°C | 40 | 19 | 14
  Fever > 39.0°C | 4 | 1 | 5
  Fever > 40.0°C | 1 | 0 | 0
  Any irratibility | 114 | 65 | 58
  Grade 2 or 3 irritability | 42 | 25 | 23
  Grade 3 irritability | 10 | 0 | 4
  Any loss of appetite | 46 | 34 | 30
  Grade 2 or 3 loss of appetite | 10 | 1 | 4
  Grade 3 loss of appetite | 1 | 0 | 0

70. Secondary Outcome: Number of Subjects Reporting Any, Grade 2 or 3 and Grade 3 Solicited General Symptoms
Description: as for outcome 69
Time Frame: Within 8 days (Day 0-7) after fourth dose vaccination
Population: The Fourth Dose Total Vaccinated cohort included all vaccinated subjects during the fourth dose phase.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 232 | 126 | 131
Participants
  Any drowsiness | 79 | 48 | 43
  Grade 2 or 3 drowsiness | 27 | 8 | 8
  Grade 3 drowsiness | 3 | 1 | 1
  Fever ≥ 38.0°C | 54 | 24 | 19
  Fever > 39.0°C | 9 | 2 | 9
  Fever > 40.0°C | 3 | 0 | 2
  Any irritability | 125 | 67 | 62
  Grade 2 or 3 irritability | 51 | 27 | 28
  Grade 3 irritability | 13 | 1 | 4
  Any loss of appetite | 56 | 35 | 33
  Grade 2 or 3 loss of appetite | 13 | 1 | 4
  Grade 3 loss of appetite | 2 | 0 | 0

71. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: as for outcome 37
Time Frame: During the 31-day follow-up period following the fourth dose
Population: The Fourth Dose Total Vaccinated cohort included all vaccinated subjects during the fourth dose phase.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 236 | 130 | 132
Participants | 102 | 39 | 58

72. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: as for outcome 38
Time Frame: as for outcome 38
Population: The Fourth Dose Total Vaccinated cohort included all vaccinated subjects during the fourth dose phase.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 236 | 130 | 132
Participants | 6 | 2 | 3

73. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Illness(es)
Description: NOCIs include autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: From receipt of the fourth dose (at Month 10-13) through the end of the 6-month safety follow-up
Population: The Fourth Dose Total Vaccinated cohort included all vaccinated subjects during the fourth dose phase.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 236 | 130 | 132
Participants | 2 | 1 | 0

74. Secondary Outcome: Number of Subjects Reporting Rash
Description: An episode of rash was defined as an episode of hives, idiopathic thrombocytopenic purpura, petechiae.
Time Frame: From receipt of the fourth dose (at Month 10-13) through the end of the 6-month safety follow-up
Population: The Fourth Dose Total Vaccinated cohort included all vaccinated subjects during the fourth dose phase.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 236 | 130 | 132
Participants | 10 | 10 | 10

75. Secondary Outcome: Number of Subjects Reporting Emergency Room (ER) Visits or Physicians Office Visits Related or Not to Common Illnesses
Description: as for outcome 42
Time Frame: From receipt of the fourth dose (at Month 10-13) through the end of the 6-month safety follow-up
Population: The Fourth Dose Total Vaccinated cohort included all vaccinated subjects during the fourth dose phase.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 236 | 130 | 132
Participants
  ER visit | 6 | 1 | 7
  Physician's office visit | 75 | 31 | 43
  Physician's o. visit not related to common illness | 13 | 8 | 13

76. Secondary Outcome: Number of Subjects Reporting Large Swelling Reactions of the Injected Limb(s)
Description: Large injection site reactions were defined as either swelling with a diameter of > 30 mm or a > 30 mm increase in the circumference of the mid-thigh when compared to the baseline (pre-vaccination) measurement, or any diffuse swelling that interfered with or prevented everyday activities (for example, active playing, eating, sleeping).
Time Frame: Within 4 days (Day 0-3) and within 8 days (Day 0-7) following the fourth dose
Population: The Fourth Dose Total Vaccinated cohort included all vaccinated subjects during the fourth dose phase.
Measure: Count of Participants; unit: Participants
Arm/Group | MenHibrix Group | ActHIB/ActHIB Group | ActHIB/MenHibrix Group
Number analyzed (Participants) | 232 | 126 | 130
Participants
  [within Day 0-3 following the fourth dose] | 3 | 0 | 0
  [within Day 0-7 following the fourth dose] | 3 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms: Within 4 or 8 days after vaccination. Unsolicited AEs: Within 31 days (Days 0-30) after vaccination. SAEs: Throughout the entire study period. Depending on groups, periods may be split into subperiods (cf below).
Description: Solicited AEs reports were not collected from Menomune Group. SAEs reporting was split: a) Day 0 to 6 months post-Dose 3 (Primary Phase groups); and b) within 31 days of 4th Dose and c) from Day 31 post 4th Dose up to 6 months afterwards (4th Dose Phase groups). N at risk for Menomune Group = N at risk for AEs occurring in at least 5% of subjects
Arm/Group | MenHibrix Group | ActHIB Group | Menomune Group | ActHIB/MenHibrix Group | ActHIB/ActHIB Group
Serious Adverse Events (participants affected / at risk) | 16/287 | 20/319 | 0/150 | 1/132 | 2/130
Other Adverse Events (participants affected / at risk) | 263/287 | 302/319 | 18/150 | 62/132 | 67/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | MenHibrix Group (N=287) | ActHIB Group (N=319) | Menomune Group (N=150) | ActHIB/MenHibrix Group (N=132) | ActHIB/ActHIB Group (N=130)
Bronchiolitis (Infections and infestations) | 4 | 5 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Dehydration (Metabolism and nutrition disorders) | 3 | 6 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Otitis media (Infections and infestations) | 3 | 1 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Viral infection (Infections and infestations) | 1 | 2 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Arachnoid cyst (Nervous system disorders) | 0 | 1 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Bronchial hyper reactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Burns first degree (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Croup infectious (Infections and infestations) | 0 | 1 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Dyskinesia (Nervous system disorders) | 0 | 1 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Erythema infectiosum (Infections and infestations) | 1 | 0 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Gastro esophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Infantile spasms (Nervous system disorders) | 0 | 1 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Influenza (Infections and infestations) | 1 | 0 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Intussusception (Gastrointestinal disorders) | 1 | 0 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Retinoblastoma bilateral (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Streptococcal bacteremia (Infections and infestations) | 1 | 0 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups
Sudden infant death syndrome (General disorders) | 1 | 0 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Tuberous sclerosis (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0/0 | 0/0 — During the entire Primary Phase of the study (study 101858), including the 6-month safety follow-up period. Groups assessed were the MenHibrix, ActHIB and Menomune groups.
Bronchiolitis (Infections and infestations) | 1/236 | 0/0 | 0/0 | 1 | 0 — During 4th Dose Phase, from the administration of Dose 4 at Month 10-13 up to Day 31 thereafter, Day 31 not included. Groups assessed were the MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups.
Abscess limb (Infections and infestations) | 0/236 | 0/0 | 0/0 | 0 | 1 — During 4th Dose Phase, from the administration of Dose 4 at Month 10-13 up to Day 31 thereafter, Day 31 not included. Groups assessed were the MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups.
Cellulitis (Infections and infestations) | 0/236 | 0/0 | 0/0 | 0 | 1 — During 4th Dose Phase, from the administration of Dose 4 at Month 10-13 up to Day 31 thereafter, Day 31 not included. Groups assessed were the MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups.
Sepsis (Infections and infestations) | 0/236 | 0/0 | 0/0 | 0 | 1 — During 4th Dose Phase, from the administration of Dose 4 at Month 10-13 up to Day 31 thereafter, Day 31 not included. Groups assessed were the MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups.
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0/236 | 0/0 | 0/0 | 1 | 0 — During 4th Dose Phase, from the administration of Dose 4 at Month 10-13 up to Day 31 thereafter, Day 31 not included. Groups assessed were the MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups.
Gastroenteritis (Infections and infestations) | 3/236 | 0/0 | 0/0 | 0 | 1 — During 4th Dose Phase, from Day 31 after administration of Dose 4up to 6 months thereafter. Groups assessed were the MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups.
Dehydration (Metabolism and nutrition disorders) | 2/236 | 0/0 | 0/0 | 0 | 0 — During 4th Dose Phase, from Day 31 after administration of Dose 4 up to 6 months thereafter. Groups assessed were the MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups.
Death (General disorders) | 1/236 | 0/0 | 0/0 | 0 | 0 — During 4th Dose Phase, from Day 31 after administration of Dose 4up to 6 months thereafter. Groups assessed were the MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups.
Febrile convulsion (Nervous system disorders) | 1/236 | 0/0 | 0/0 | 0 | 0 — During 4th Dose Phase, from Day 31 after administration of Dose 4 up to 6 months thereafter. Groups assessed were the MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups.
Hypoglycemia (Metabolism and nutrition disorders) | 0/236 | 0/0 | 0/0 | 1 | 0 — During 4th Dose Phase, from Day 31 after administration of Dose 4up to 6 months thereafter. Groups assessed were the MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups.
Hypokalemia (Metabolism and nutrition disorders) | 1/236 | 0/0 | 0/0 | 0 | 0 — During 4th Dose Phase, from Day 31 after administration of Dose 4up to 6 months thereafter. Groups assessed were the MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups.
Respiratory syncytial virus infection (Infections and infestations) | 0/236 | 0/0 | 0/0 | 0 | 1 — During 4th Dose Phase, from Day 31 after administration of Dose 4 up to 6 months thereafter. Groups assessed were the MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | MenHibrix Group (N=287) | ActHIB Group (N=319) | Menomune Group (N=150) | ActHIB/MenHibrix Group (N=132) | ActHIB/ActHIB Group (N=130)
Pain (General disorders) | 129/286 | 171/317 | 0/0 | 0/0 | 0/0 — During Primary Phase (study 101858), within the 4 days following primary vaccination course. Primary Phase solicited symptoms reports were collected from the MenHibrix and ActHIB groups only, solely from subjects with data available.
Redness (General disorders) | 112/286 | 148/317 | 0/0 | 0/0 | 0/0 — During Primary Phase (study 101858), within the 4 days following primary vaccination course. Primary Phase solicited symptoms reports were collected from the MenHibrix and ActHIB groups only, solely from subjects with data available.
Swelling (General disorders) | 90/286 | 110/317 | 0/0 | 0/0 | 0/0 — During Primary Phase (study 101858), within the 4 days following primary vaccination course. Primary Phase solicited symptoms reports were collected from the MenHibrix and ActHIB groups only, solely from subjects with data available.
Pain (General disorders) | 129/286 | 171/317 | 0/0 | 0/0 | 0/0 — During Primary Phase (study 101858), within the 8 days following primary vaccination course. Primary Phase solicited symptoms reports were collected from the MenHibrix and ActHIB groups only, solely from subjects with data available.
Redness (General disorders) | 113/286 | 148/317 | 0/0 | 0/0 | 0/0 — During Primary Phase (study 101858), within the 8 days following primary vaccination course. Primary Phase solicited symptoms reports were collected from the MenHibrix and ActHIB groups only, solely from subjects with data available.
Swelling (General disorders) | 90/286 | 111/317 | 0/0 | 0/0 | 0/0 — During Primary Phase (study 101858), within the 8 days following primary vaccination course. Primary Phase solicited symptoms reports were collected from the MenHibrix and ActHIB groups only, solely from subjects with data available.
Drowsiness (General disorders) | 185/286 | 224/317 | 0/0 | 0/0 | 0/0 — During Primary Phase (study 101858), within the 4 days following primary vaccination course. Primary Phase solicited symptoms reports were collected from the MenHibrix and ActHIB groups only, solely from subjects with data available.
Fever (General disorders) | 110/286 | 150/317 | 0/0 | 0/0 | 0/0 — During Primary Phase (study 101858), within the 4 days following primary vaccination course. Primary Phase solicited symptoms reports were collected from the MenHibrix and ActHIB groups only, solely from subjects with data available.
Irritability (General disorders) | 217/286 | 268/317 | 0/0 | 0/0 | 0/0 — During Primary Phase (study 101858), within the 4 days following primary vaccination course. Primary Phase solicited symptoms reports were collected from the MenHibrix and ActHIB groups only, solely from subjects with data available.
Loss of appetite (General disorders) | 123/286 | 159/317 | 0/0 | 0/0 | 0/0 — During Primary Phase (study 101858), within the 4 days following primary vaccination course. Primary Phase solicited symptoms reports were collected from the MenHibrix and ActHIB groups only, solely from subjects with data available.
Drowsiness (General disorders) | 187/286 | 227/317 | 0/0 | 0/0 | 0/0 — During Primary Phase (study 101858), within the 8 days following primary vaccination course. Primary Phase solicited symptoms reports were collected from the MenHibrix and ActHIB groups only, solely from subjects with data available.
Fever (General disorders) | 115/286 | 158/317 | 0/0 | 0/0 | 0/0 — During Primary Phase (study 101858), within the 8 days following primary vaccination course. Primary Phase solicited symptoms reports were collected from the MenHibrix and ActHIB groups only, solely from subjects with data available.
Irritability (General disorders) | 222/286 | 272/317 | 0/0 | 0/0 | 0/0 — During Primary Phase (study 101858), within the 8 days following primary vaccination course. Primary Phase solicited symptoms reports were collected from the MenHibrix and ActHIB groups only, solely from subjects with data available.
Loss of appetite (General disorders) | 127/286 | 164/317 | 0/0 | 0/0 | 0/0 — During Primary Phase (study 101858), within the 8 days following primary vaccination course. Primary Phase solicited symptoms reports were collected from the MenHibrix and ActHIB groups only, solely from subjects with data available.
Upper respiratory tract infection (Infections and infestations) | 77 | 71 | 4 | 0/0 | 0/0 — Unsolicited AE reported during Primary Phase (study 101858), within the 31-day follow-up period after primary vaccination course. Group assessed for unsolicited AEs during that period were the MenHibrix, ActHIB and Menomune groups
Otitis media (Infections and infestations) | 67 | 55 | 6 | 0/0 | 0/0 — Unsolicited AE reported during Primary Phase (study 101858), within the 31-day follow-up period after primary vaccination course. Group assessed for unsolicited AEs during that period were the MenHibrix, ActHIB and Menomune groups
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 29 | 18 | 3 | 0/0 | 0/0 — Unsolicited AE reported during Primary Phase (study 101858), within the 31-day follow-up period after primary vaccination course. Group assessed for unsolicited AEs during that period were the MenHibrix, ActHIB and Menomune groups
Bronchiolitis (Infections and infestations) | 21 | 25 | 0 | 0/0 | 0/0 — Unsolicited AE reported during Primary Phase (study 101858), within the 31-day follow-up period after primary vaccination course. Group assessed for unsolicited AEs during that period were the MenHibrix, ActHIB and Menomune groups
Viral infection (Infections and infestations) | 15 | 21 | 2 | 0/0 | 0/0 — Unsolicited AE reported during Primary Phase (study 101858), within the 31-day follow-up period after primary vaccination course. Group assessed for unsolicited AEs during that period were the MenHibrix, ActHIB and Menomune groups
Eczema (Skin and subcutaneous tissue disorders) | 13 | 23 | 0 | 0/0 | 0/0 — Unsolicited AE reported during Primary Phase (study 101858), within the 31-day follow-up period after primary vaccination course. Group assessed for unsolicited AEs during that period were the MenHibrix, ActHIB and Menomune groups
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 18 | 4 | 0/0 | 0/0 — Unsolicited AE reported during Primary Phase (study 101858), within the 31-day follow-up period after primary vaccination course. Group assessed for unsolicited AEs during that period were the MenHibrix, ActHIB and Menomune groups
Conjunctivitis (Eye disorders) | 11 | 21 | 0 | 0/0 | 0/0 — Unsolicited AE reported during Primary Phase (study 101858), within the 31-day (Days 0-30) follow-up period after primary vaccination course. Group assessed for unsolicited AEs during that period were the MenHibrix, ActHIB and Menomune groups.
Diarrhea (Gastrointestinal disorders) | 15 | 16 | 1 | 0/0 | 0/0 — Unsolicited AE reported during Primary Phase (study 101858), within the 31-day (Days 0-30) follow-up period after primary vaccination course. Group assessed for unsolicited AEs during that period were the MenHibrix, ActHIB and Menomune groups.
Flatulence (Gastrointestinal disorders) | 16 | 7 | 0 | 0/0 | 0/0 — Unsolicited AE reported during Primary Phase (study 101858), within the 31-day (Days 0-30) follow-up period after primary vaccination course. Group assessed for unsolicited AEs during that period were the MenHibrix, ActHIB and Menomune groups.
Limb circumference (General disorders) | 59/232 | 0/0 | 0/0 | 36/130 | 44/126 — During 4th Dose Phase (study 102015), within the 4 days after 4th dose vaccination. Symptom reports were collected from all groups in this phase (MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups), from subjects with data available.
Pain (General disorders) | 79/232 | 0/0 | 0/0 | 48/130 | 42/126 — During 4th Dose Phase (study 102015), within the 8 days after 4th dose vaccination. Symptom reports were collected from all groups in this phase (MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups), solely from subjects with data available.
Redness (General disorders) | 81/232 | 0/0 | 0/0 | 38/130 | 40/126 — During 4th Dose Phase (study 102015), within the 8 days after 4th dose vaccination. Symptom reports were collected from all groups in this phase (MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups), solely from subjects with data available.
Swelling (General disorders) | 49/232 | 0/0 | 0/0 | 20/130 | 19/126 — During 4th Dose Phase (study 102015), within the 8 days after 4th dose vaccination. Symptom reports were collected from all groups in this phase (MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups), from subjects with data available.
Drowsiness (General disorders) | 72/232 | 0/0 | 0/0 | 41/131 | 48/126 — During 4th Dose Phase (study 102015), within the 8 days after 4th dose vaccination. Symptom reports were collected from all groups in this phase (MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups), from subjects with data available.
Fever (General disorders) | 40/232 | 0/0 | 0/0 | 14/131 | 19/126 — During 4th Dose Phase (study 102015), within the 4 days after 4th dose vaccination. Symptom reports were collected from all groups in this phase (MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups), from subjects with data available.
Irritability (General disorders) | 114/232 | 0/0 | 0/0 | 58/131 | 65/126 — During 4th Dose Phase (study 102015), within the 8 days after 4th dose vaccination. Symptom reports were collected from all groups in this phase (MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups), from subjects with data available.
Loss of appetite (General disorders) | 46/232 | 0/0 | 0/0 | 30/131 | 34/126 — During 4th Dose Phase (study 102015), within the 8 days after 4th dose vaccination. Symptom reports were collected from all groups in this phase (MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups), from subjects with data available.
Limb circumference (General disorders) | 61/232 | 0/0 | 0/0 | 36/130 | 46/126 — During 4th Dose Phase (study 102015), within the 4 days after 4th dose vaccination. Symptom reports were collected from all groups in this phase (MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups), from subjects with data available.
Pain (General disorders) | 79/232 | 0/0 | 0/0 | 48/130 | 42/126 — During 4th Dose Phase (study 102015), within the 4 days after 4th dose vaccination. Symptom reports were collected from all groups in this phase (MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups), from subjects with data available.
Redness (General disorders) | 81/232 | 0/0 | 0/0 | 39/130 | 40/126 — During 4th Dose Phase (study 102015), within the 4 days after 4th dose vaccination. Symptom reports were collected from all groups in this phase (MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups), from subjects with data available.
Swelling (General disorders) | 49/232 | 0/0 | 0/0 | 20/130 | 19/126 — During 4th Dose Phase (study 102015), within the 4 days after 4th dose vaccination. Symptom reports were collected from all groups in this phase (MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups), from subjects with data available.
Drowsiness (General disorders) | 79/232 | 0/0 | 0/0 | 43/131 | 48/126 — During 4th Dose Phase (study 102015), within the 4 days after 4th dose vaccination. Symptom reports were collected from all groups in this phase (MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups), from subjects with data available.
Fever (General disorders) | 54/232 | 0/0 | 0/0 | 19/131 | 24/126 — During 4th Dose Phase (study 102015), within the 4 days after 4th dose vaccination. Symptom reports were collected from all groups in this phase (MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups), from subjects with data available.
Irritability (General disorders) | 125/232 | 0/0 | 0/0 | 62/131 | 67/126 — During 4th Dose Phase (study 102015), within the 4 days after 4th dose vaccination. Symptom reports were collected from all groups in this phase (MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups), from subjects with data available.
Loss of appetite (General disorders) | 56/232 | 0/0 | 0/0 | 33/131 | 35/126 — During 4th Dose Phase (study 102015), within the 4 days after 4th dose vaccination. Symptom reports were collected from all groups in this phase (MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups), from subjects with data available.
Otitis media (Infections and infestations) | 26/236 | 0/0 | 0/0 | 12 | 11 — Unsolicited AE reported during 4th Dose Phase (study 102015), within the 31-day follow-up period after 4th-dose vaccination. Group assessed for unsolicited AEs during that period were the MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups
Upper respiratory tract infection (Infections and infestations) | 22/236 | 0/0 | 0/0 | 5 | 10 — Unsolicited AE reported during 4th Dose Phase (study 102015), within the 31-day follow-up period after 4th-dose vaccination. Group assessed for unsolicited AEs during that period were the MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups
Teething (Gastrointestinal disorders) | 19/236 | 0/0 | 0/0 | 5 | 3 — Unsolicited AE reported during 4th Dose Phase (study 102015), within the 31-day follow-up period after 4th-dose vaccination. Group assessed for unsolicited AEs during that period were the MenHibrix, ActHIB/ActHIB and ActHIB/MenHibrix groups

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.